CLINICAL TRIAL: NCT01324284
Title: Comparative Study of Lubiprostone and PEG Preparation Versus Conventional PEG Preparation to Enhance the Colonoscopy Preparation Quality in an Indian Tertiary Care Center.
Brief Title: Comparative Study of Lubiprostone and PEG Preparation Versus Conventional PEG Preparation for Colonoscopy
Acronym: Lubiprostone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Rupa Banerjee, Consultant gastroenterologist, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: AIG-GI2011-01
Record Dates: First submitted 2011-03-22; First posted 2011-03-29 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Colorectal Carcinoma
Keywords: Lubiprostone; Bowel preparation regime
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Lubiprostone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lubiprostone (Experimental): Lubiprostone with PEG solution versus Placebo with PEG solution
  Interventions: Drug: Lubiprostone
- lubiprostone versus placebo (Placebo Comparator)

INTERVENTIONS:
Drug: Lubiprostone — Lubiprostone is a chloride channel activator approved by the Food and Drug Administration for the treatment of chronic constipation. A randomized, double-blind, parallel-group, placebo-controlled study evaluating the effect of lubiprostone on gastric function showed slowed gastric emptying and increased small bowel and colonic transit time. Peak plasma concentration was shown to be around 1.14 hours, with a majority of the drug excreted in the urine within 48 hours.
  Arms: Lubiprostone

SUMMARY:
Lubiprostone as an adjunct to the standard bowel preparation regime the quality of bowel preparation can be improved for a good colonoscopic examination without missing lesions and complications.

DETAILED DESCRIPTION:
Objectives:

1. Primary:

   * Same day Low volume PEG with placebo (Arm 1) versus same day low volume PEG with Lubiprostone (Arm 2)
   * Waiting time for colonoscopic procedure and quality of bowel preparation
2. Secondary:

   * Quality of bowel preparation without Dietary restriction (Modified bowel preparation regime without Fiber diet restrictions)

ELIGIBILITY:
Inclusion Criteria:

1. All adult patient referred for colonoscopy to AIG
2. Age 18 - 75 years old

Exclusion Criteria:

1. Acute GI bleeding.
2. Patient of bowel preparation regime other than excepted for the study.
3. Renal insufficiency.
4. Dementia.
5. Symptomatic heart failure.
6. Recent Myocardial Infarction.
7. Patients with ileus.
8. Suspected bowel obstruction.
9. Prior alimentary tract surgery.
10. Significant gastroparesis.
11. Gastric outlet obstruction.
12. Toxic colitis or megacolon.
13. Pregnant or lactating patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Quality of bowel preparation in Same day Low volume PEG with placebo versus same day low volume PEG with Lubiprostone | 2 months
  Quality of bowel preparation is based on Boston Bowel Preparation Score (BBPS)

CONTACTS AND LOCATIONS:
Overall Officials: Nageshwar D Reddy, MD. DM, Study Director — Asian Institute of Gastroenterolgy India; Rupa Banerjee, MD, Principal Investigator — Asian Institute of Gastroenterology, India; Saravanan Arjunan, MD, Principal Investigator — Asian Institute of Gastroenterology, India; Manu Tandan, MD DM, Principal Investigator — AIG Hyderabad india

REFERENCES:
- [Derived] Banerjee R, Chaudhari H, Shah N, Saravanan A, Tandan M, Reddy DN. Addition of Lubiprostone to polyethylene glycol(PEG) enhances the quality & efficacy of colonoscopy preparation: a randomized, double-blind, placebo controlled trial. BMC Gastroenterol. 2016 Oct 13;16(1):133. doi: 10.1186/s12876-016-0542-0. PMID 27737636